CLINICAL TRIAL: NCT04155723
Title: Impact of a Task Delegation to ICU Nurses for Midlines' Placement on the Duration of Exposure to Central Venous Catheters
Brief Title: Impact of a Task Delegation to ICU Nurses for Midlines' Placement
Acronym: IDEM
Status: Completed | Type: Observational
Sponsor: Groupe Hospitalier de Bretagne Sud (Other)
Responsible Party: Principal Investigator, Pierre Bouju, Principal Investigator, Groupe Hospitalier de Bretagne Sud
Other Study IDs: GHBretagneSud
Record Dates: First submitted 2019-10-25; First posted 2019-11-07 (Actual); Last update posted 2023-07-12 (Actual); Status verified 2023-07

CONDITIONS: Catheter-Related Infections
Keywords: Midlines
MeSH Terms: conditions — Catheter-Related Infections

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Phase 1 group: During phase 1, Midlines are inserted only by doctors.
- Phase 2 group: During Phase 2, Midlines are preferentially inserted by ICU nurses, and if needed, by doctors.

SUMMARY:
The administration of medication, fluid resuscitation, or even nutrition in intensive care unit (ICU) patients, requires one or more infusion lines which can be peripheral or central. Midline catheter is a 10 to 20 cm long peripheral venous catheter, which can be used for up to 28 days. These features make it a good alternative to central venous and conventional peripheral venous catheters.

Midlines are routinely used in the ICU of Lorient Hospital, currently inserted by doctors. In association with the Regional Health Agency, the investigators are currently implementing a project of task delegation to ICU nurses, so that they could insert Midlines' catheters. The aim of the study is to increase the use of Midlines in the unit to reduce the exposure to central venous catheters and their complications, such as infections or thrombosis.

The investigators propose to conduct a prospective monocentric study to compare the frequency of Midlines'use, before and after the task delegation. The primary objective is to compare the duration of exposure to central venous catheters between the two periods. Secondary objectives are to compare the duration of exposure to peripheral venous catheters and Midlines, and the catheter-related infections and thrombosis.

DETAILED DESCRIPTION:
The administration of medication, fluid resuscitation, or even nutrition in intensive care unit (ICU) patients, requires one or more infusion lines which can be peripheral or central. Although central venous catheters (CVC) are often mandatory in ICU, the risk of catheter-related infections should lead to consider the insertion of peripheral venous catheters. However in ICU patients, presence of edema or poor venous condition may not allow placement of peripheral venous catheter.

Midline catheter is a 10 to 20 cm long peripheral venous catheter, which can be used for up to 28 days (according to manufacturer recommendations). These features make it a good alternative to central venous and conventional peripheral venous catheters. They are placed at the bedside, peripherally into the cephalic or basilic vein, with the tip reaching the axillary vein.

Midlines are routinely used in the ICU of Lorient Hospital, currently inserted by doctors. Studies have shown the feasibility and the safety of delegating to nurses placement of CVC and Midlines. In association with the Regional Health Agency, the investigators are currently implementing a project of task delegation to ICU nurses, so that they could insert Midlines' catheters.

Midlines' implementation has been associated with a decrease in the use of CVC and catheter-related infections. To our knowledge, no study investigated the placement of Midlines by nurses in the ICU.

The investigators propose to conduct a prospective monocentric study to compare the frequency of Midlines' use, before and after the task delegation. The primary objective is to compare the duration of exposure to central venous catheters between the two periods. Secondary objectives are to compare the duration of exposure to peripheral venous catheters and Midlines, and the catheter-related infections and thrombosis. Complications related to Midlines' placement would also be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients hospitalized in ICU for more than 48 hours

Exclusion Criteria:

* Patient under 18 years old
* Patient under legal guardianship
* Absence of health insurance in France
* Refusal of the patient or his next-of-kin
* Patient with a decision of withholding or withdrawing of life sustaining therapy
* Patient with a subcutaneous central venous port
* Impossibility of infusion on the upper limbs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients hospitalized in ICU for more than 48 hours
Sampling Method: Non-Probability Sample
Enrollment: 310 (Actual)
Dates: Start 2019-11-06 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
Duration of exposure to central venous catheter | ICU discharge (usually seven days)
  Duration of exposure to central venous catheter (catheter-days per patient-day)

SECONDARY OUTCOMES:
Duration of exposure to peripheral venous catheter | ICU discharge (usually seven days)
  Duration of exposure to peripheral venous catheter (catheter-days per patient-day)
Duration of exposure to Midline | ICU discharge (usually seven days)
  Duration of exposure to Midline (catheter-days per patient-day)
Number of catheter-related infections | ICU discharge (usually seven days)
  Number of catheter-related infections (number of events per 1000 catheter days)
Number of catheter-related infections | Hospital discharge (usually two weeks)
  Number of catheter-related infections (number of events per 1000 catheter days)
Number of catheter-related thrombosis | ICU discharge (usually seven days)
  Number of catheter-related thrombosis (number of events per 1000 catheter days)
Number of catheter-related thrombosis | Hospital discharge (usually two weeks)
  Number of catheter-related thrombosis (number of events per 1000 catheter days)
Number of pneumothorax and arterial punctures | ICU discharge (usually seven days)
  Number of pneumothorax and arterial punctures (for each catheter inserted, percentage)
Number of patients discharged from the ICU with a central venous catheter | ICU discharge (usually seven days)
  Number of patients discharged from the ICU with a central venous catheter (percentage)
Description of the events associated with Midlines' insertion : Number of punctures | ICU discharge (usually seven days)
  Number of punctures (per Midline inserted)
Description of the events associated with Midlines' insertion : Duration of the procedure | ICU discharge (usually seven days)
  Duration of the procedure (in minutes)
Description of the events associated with Midlines' insertion : Failure rate | ICU discharge (usually seven days)
  Failure rate (percentage)

CONTACTS AND LOCATIONS:
Locations (1):
- Groupe Hospitalier Bretagne Sud, Lorient, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] O'Grady NP, Alexander M, Burns LA, Dellinger EP, Garland J, Heard SO, Lipsett PA, Masur H, Mermel LA, Pearson ML, Raad II, Randolph AG, Rupp ME, Saint S; Healthcare Infection Control Practices Advisory Committee. Guidelines for the prevention of intravascular catheter-related infections. Am J Infect Control. 2011 May;39(4 Suppl 1):S1-34. doi: 10.1016/j.ajic.2011.01.003. No abstract available. PMID 21511081
- [Background] Pathak R, Patel A, Enuh H, Adekunle O, Shrisgantharajah V, Diaz K. The Incidence of Central Line-Associated Bacteremia After the Introduction of Midline Catheters in a Ventilator Unit Population. Infect Dis Clin Pract (Baltim Md). 2015 May;23(3):131-134. doi: 10.1097/IPC.0000000000000237. PMID 25972725
- [Background] Pathak R, Gangina S, Jairam F, Hinton K. A vascular access and midlines program can decrease hospital-acquired central line-associated bloodstream infections and cost to a community-based hospital. Ther Clin Risk Manag. 2018 Aug 21;14:1453-1456. doi: 10.2147/TCRM.S171748. eCollection 2018. PMID 30174427
- [Background] Xu T, Kingsley L, DiNucci S, Messer G, Jeong JH, Morgan B, Shutt K, Yassin MH. Safety and utilization of peripherally inserted central catheters versus midline catheters at a large academic medical center. Am J Infect Control. 2016 Dec 1;44(12):1458-1461. doi: 10.1016/j.ajic.2016.09.010. PMID 27908432
- [Background] Shokoohi H, Boniface K, McCarthy M, Khedir Al-tiae T, Sattarian M, Ding R, Liu YT, Pourmand A, Schoenfeld E, Scott J, Shesser R, Yadav K. Ultrasound-guided peripheral intravenous access program is associated with a marked reduction in central venous catheter use in noncritically ill emergency department patients. Ann Emerg Med. 2013 Feb;61(2):198-203. doi: 10.1016/j.annemergmed.2012.09.016. Epub 2012 Nov 7. PMID 23141920
- [Background] Alexandrou E, Spencer TR, Frost SA, Mifflin N, Davidson PM, Hillman KM. Central venous catheter placement by advanced practice nurses demonstrates low procedural complication and infection rates--a report from 13 years of service*. Crit Care Med. 2014 Mar;42(3):536-43. doi: 10.1097/CCM.0b013e3182a667f0. PMID 24145843